CLINICAL TRIAL: NCT02228057
Title: Long Term Patency Following Arterial Repair
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Alexander M Spiess, MD, Dr., University of Pittsburgh
Other Study IDs: PRO12010024
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Upper Extremity Arterial Surgery
Keywords: arterial patency; upper extremity; anastomosis; sensibility; pain; cold intolerance
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- operated group: all patients who had upper extremity artery surgery at least 6 months ago

SUMMARY:
Injury to the blood vessels of the extremities, and more specifically the arteries, can result from fractures and severe crush injuries. It occurs in about 3% of the general population. People affected by blood vessel injuries can have important problems, including cold intolerance, general pain, and weakened function of the associated limb. Even after surgical intervention to repair the affected artery, people may still experience numbness, problems with movement, and an inadequate supply of oxygen to the limb. These symptoms are particularly relevant in the case of forearm arterial repairs because this repair directly affects one of our most vital structures: the hand. Despite available interventions and advances in microsurgical technique, arterial repairs can still result in significant sensory and functional impairment of the hand. Once an artery within the arm is injured, a surgeon's primary goal is to restore blood flow to the hand and prevent functional impairment. Even with a prompt effort to restore hand perfusion, long-term (greater than 6 months) sensory and motor function is hard to predict.

Furthermore, sometimes the repaired artery becomes occluded over time. We believe that this occlusion has a direct impact on a patient's perceived pain and cold intolerance at the level of the hand.

In this study, we are investigating the occurrence of blood vessel occlusion in the arm after at least 6 months of surgery and the impact of this event. To assess this we will use physical exams, non-invasive tests, duplex doppler ultrasound and questionnaires. Questionnaires, including the DASH (disabilities of the arm, shoulder,and hand), CISS (Cold Intolerance Symptom Severity Questionnaire), and Michigan hand score, will be used to assess pain, sensory, and motor impairments in both the affected and unaffected hand. Functional assessments will include 2-point discrimination, grip strength, pinch strength, capillary refill and range of motion.

DETAILED DESCRIPTION:
Vascular injuries of the extremities can result from fractures, severe crush injuries, lacerations, and even iatrogenic causes, such as surgical interventions. Its prevalence is about 3% in the general population with increased incidence during times of war. Patients affected by vascular injuries can have significant morbidities, including cold intolerance, pain, sensory abnormalities, and weakness of the affected limb. Even after repair of the affected artery, patients may still experience paresthesias, motor function abnormalities and pain and cold intolerance. These symptoms are particularly relevant in the case of arm arterial repairs because this repair directly affects the function of the hand. Different techniques of arterial repair have evolved over time. Venous grafts (i.e. saphenous and dorsal hand veins) can be employed to repair the damaged vessel. Although most appropriate for treating long gaps, vein grafts have several disadvantages. There is often a diameter mismatch between the harvested vein and the damaged artery which can compromise the repair site. Furthermore, veins are more compliant and have higher volume storage capabilities than their arterial counterparts. These inherent venous qualities can alter blood flow to the limb causing stasis, turbulence, and eventually, stenosis of the graft. Other methodologies have been developed in an effort to balance the negatives associated with venous grafting, including synthetic graft use, arterial ligation, end-to-side anastomosis, and end-to-end repair. Despite available interventions and advances in microsurgical technique, arterial repair in the arm, can still result in significant functional impairment of the upper extremity. The hand is highly perfused with a dual arterial system that arches across the dorsal and palmar surface of the hand. Once an upper extremity artery is compromised, a surgeon's primary goal is to restore blood flow to the hand so as to prevent impairment. Despite a surgeon's best efforts, long term (greater than 6 months) outcomes are hard to predict. Furthermore, the patency rates of the arterial repair have been consistently reported at approximately 50%. We believe that the long term patency of the upper extremity artery has a direct effect on a patient's perceived pain and cold intolerance, sensibility, and motor function of the hand. Our hypothesis is that repaired arteries in the upper extremity will have an occlusion rate of 50% in the long term (greater than 6 months post-surgery) and that this occlusion is responsible for motor and sensory function abnormalities, pain, and cold-intolerance. We will use high resolution duplex Doppler ultrasound to investigate occlusion rates of repaired arteries and compare those to the unaffected contralateral arteries (internal control). Questionnaires, including the DASH (disabilities of the arm, shoulder, and hand), CISS (Cold Intolerance Symptom Severity Questionnaire), and Michigan hand score, will be used to assess pain, cold intolerance, sensory, and motor impairments in both the affected and unaffected hand. Functional assessments will include 2-point discrimination, grip strength, pinch strength, capillary refill and range of motion.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting the following criteria will be eligible to participate in this study:

1. Age 18 and over
2. Able to provide informed consent
3. Have previously underwent surgery for an arm arterial repair
4. Be at least 6 months post-arterial repair
5. Willing and able to comply with follow-up tests/procedures and questionnaires

Exclusion Criteria:

Patients meeting the following criteria will be excluded from this study:

1. Age less than 18 years
2. Unable to provide informed consent
3. Nerve repair in extremity of interest
4. Any condition which compromises the contralateral hand to serve as a reliable internal control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients that underwent upper extremity arterial surgery and are at least 6 months out of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
relationship of time after arterial repair with patency of the vessel | at least 6 months after surgery
  By using ultrasound, both the ulnar and radial artery will be visualized in both arms and using color ultrasound, we will detect the bloodflow. If no flow is present we will assume that the vessel is occluded.

SECONDARY OUTCOMES:
Correlation between arterial patency and cold intolerance. | at least 6 months after surgery
  Both hands will be assessed for cold intolerance. To assess this we will use the CISS questionnaire (Cold Intolerance Symptom Severity Questionnaire).
Correlation between arterial patency and digital sensibility. | at least 6 months after surgery
  Both hands will be assessed for sensibility. To assess this we will use physical exams and questionnaires. Questionnaires, including the DASH (disabilities of the arm, shoulder,and hand) and Michigan hand score will be used to assess sensibility in both the affected and unaffected hand. A functional assessment for sensibility will be the 2-point discrimination.
Correlation between arterial patency and hand strength. | at least 6 months after surgery
  Functional assessments will include grip strength and pinch strength.
Correlation between arterial patency and capillary refill | at least 6 months after surgery
  Vascular assessment will include capillary refill.
Correlation between arterial patency and range of movement of the fingers | at least 6 months after surgery
  Functional assessments will include the measurement of the distance of the fingertips to the distal palmar crease when the fingers are maximally flexed.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander M. Spiess, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Scaife Hall, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Knobloch K, Vogt PM. On "patency of radial arteries reconstructed after radial forearm flap harvest (J Reconstr Microsurg 2007;23:347-350)". J Reconstr Microsurg. 2009 Jan;25(1):77-8; author reply 79-80. doi: 10.1055/s-0028-1090602. Epub 2008 Oct 16. No abstract available. PMID 18925541
- [Background] Gelberman RH, Nunley JA, Koman LA, Gould JS, Hergenroeder PT, MacClean CR, Urbaniak JR. The results of radial and ulnar arterial repair in the forearm. Experience in three medical centers. J Bone Joint Surg Am. 1982 Mar;64(3):383-7. PMID 7061556
- [Background] Nunley JA, Goldner RD, Koman LA, Gelberman R, Urbaniak JR. Arterial stump pressure: a determinant of arterial patency? J Hand Surg Am. 1987 Mar;12(2):245-9. doi: 10.1016/s0363-5023(87)80280-0. PMID 3559079
- [Background] Lee RE, Obeid FN, Horst HM, Bivins BA. Acute penetrating arterial injuries of the forearm. Ligation or repair? Am Surg. 1985 Jun;51(6):318-24. PMID 3994174
- [Background] Deutinger M, Porenta G, Metz V, Kaliman J, Freilinger G. [Hemodynamic and clinical studies following injury of the arteries of the forearm]. Handchir Mikrochir Plast Chir. 1989 Nov;21(6):283-6. German. PMID 2606367
- [Background] Aftabuddin M, Islam N, Jafar MA, Haque E, Alimuzzaman M. Management of isolated radial or ulnar arteries at the forearm. J Trauma. 1995 Jan;38(1):149-51. doi: 10.1097/00005373-199501000-00033. PMID 7745646
- [Background] Daoutis N, Gerostathopoulos N, Bouchlis G, Efstathopoulos D, Misitzis D, Anagnostou S, Vasiliadiw A. Results after repair of traumatic arterial damage in the forearm. Microsurgery. 1992;13(4):175-7. doi: 10.1002/micr.1920130405. PMID 1495376
- [Background] Johnson M, Ford M, Johansen K. Radial or ulnar artery laceration. Repair or ligate? Arch Surg. 1993 Sep;128(9):971-4; discussion 974-5. doi: 10.1001/archsurg.1993.01420210031004. PMID 8368933
- [Background] Ge XZ, Huang GK. Use of distal arteries for microvascular reconstruction in forearm and hand surgery. Microsurgery. 1996;17(4):180-3. doi: 10.1002/(SICI)1098-2752(1996)17:43.0.CO;2-P. PMID 9140949
- [Background] Hentschel M, Rucker G. [Treatment of arterial injuries of the forearm and hand]. Handchirurgie. 1970;2(1):18-21. No abstract available. German. PMID 5538419
- [Background] Stricker SJ, Burkhalter WE, Ouellette AE. Single-vessel forearm arterial repairs. Patency rates using nuclear angiography. Orthopedics. 1989 Jul;12(7):963-5. doi: 10.3928/0147-7447-19890701-08. PMID 2771822
- [Background] Gelberman RH, Blasingame JP, Fronek A, Dimick MP. Forearm arterial injuries. J Hand Surg Am. 1979 Sep;4(5):401-8. doi: 10.1016/s0363-5023(79)80031-3. PMID 501048
- [Background] Rothkopf DM, Chu B, Gonzalez F, Borah G, Ashmead D 4th, Dunn R. Radial and ulnar artery repairs: assessing patency rates with color Doppler ultrasonographic imaging. J Hand Surg Am. 1993 Jul;18(4):626-8. doi: 10.1016/0363-5023(93)90305-M. PMID 8349969